CLINICAL TRIAL: NCT06771609
Title: Evaluate the Efficacy and Safety of PD-L1 Monoclonal Antibody Combined with VEX Metronomic Chemotherapy with or Without Radiotherapy in Advanced Triple-negative Breast Cancer: a Prospective, Multicenter, Randomized Controlled Phase II Clinical Trial.
Brief Title: Phase II Clinical Trial of PD-L1 in Combination with Vinorelbine + Cyclophosphamide + Capecitabine (VEX) Metronomic Chemotherapy with or Without Radiotherapy for Advanced Triple-negative Breast Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Deputy Director of the Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC4907
Record Dates: First submitted 2024-12-10; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-09

CONDITIONS: Advanced Triple-negative Breast Cancer
Keywords: advanced triple-negative breast cancer; PD-L1 in combination with VEX metronomic chemotherapy; radiotherapy
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adebry single antibody + VEX metronomic chemotherapy + radiotherapy (Experimental): 1. Adebry antibody: 1200mg on day 1, every 3 weeks；
  2. vinorelbine + cyclophosphamide + capecitabine (VEX) metronomic chemotherapy: Vinorelbine 20mg orally, once every other day, Q3W Cyclophosphamide 50mg orally, once daily, Q3W Capecitabine 500mg orally, three times daily, Q3W
  3. Radiotherapy: Radiotherapy is administered within 3 weeks after the first immunotherapy. Different radiotherapy techniques are chosen based on the size and location of the metastatic lesions: Stereotactic Body Radiation Therapy (SBRT), Spatially Fractionated Radiation Therapy (SFRT), or Low-dose Radiotherapy (LDRT).
  Interventions: Drug: Adebry single antibody + VEX metronomic chemotherapy + radiotherapy
- debry single antibody + VEX metronomic chemotherapy (Active Comparator): 1. Adebry antibody: 1200mg on day 1, every 3 weeks；
  2. VEX Metronomic Chemotherapy:
  Vinorelbine 20mg orally, once every other day, Q3W Cyclophosphamide 50mg orally, once daily, Q3W Capecitabine 500mg orally, three times daily, Q3W
  Interventions: Drug: debry single antibody + VEX metronomic chemotherapy

INTERVENTIONS:
Drug: Adebry single antibody + VEX metronomic chemotherapy + radiotherapy — 1、Adebry antibody: 1200mg on day 1, every 3 weeks； 2、VEX Metronomic Chemotherapy: Vinorelbine 20mg orally, once every other day, Q3W Cyclophosphamide 50mg orally, once daily, Q3W Capecitabine 500mg orally, three times daily, Q3W
  Arms: Adebry single antibody + VEX metronomic chemotherapy + radiotherapy
Drug: debry single antibody + VEX metronomic chemotherapy — 1、Adebry antibody: 1200mg on day 1, every 3 weeks； 2、VEX Metronomic Chemotherapy: Vinorelbine 20mg orally, once every other day, Q3W Cyclophosphamide 50mg orally, once daily, Q3W Capecitabine 500mg orally, three times daily, Q3W
  Arms: debry single antibody + VEX metronomic chemotherapy

SUMMARY:
Phase II clinical trial of PD-L1 in combination with vinorelbine + cyclophosphamide + capecitabine (VEX) metronomic chemotherapy with or without radiotherapy for advanced triple-negative breast cancer.

ELIGIBILITY:
Subjects are eligible to be included in the study only if all of the following criteria apply:

1. Male or female who is 18 years of age or older on the day of signing the informed consent form.
2. Subjects with metastatic triple-negative breast cancer, with clear clinical data records; specific reference to the "American Society of Clinical Oncology - College of American Pathologists (ASCO/CAP) guidelines."
3. Have received less than or equal to 1 line of chemotherapy for metastatic breast cancer;
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 as assessed within 10 days before the start of study treatment;
5. Subjects must have at least one measurable lesion present; specific reference to the "Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)" guidelines;
6. Subjects may have previously received treatment with anthracyclines (e.g., doxorubicin, epirubicin) and/or taxanes (e.g., paclitaxel, docetaxel) as follows: a) The subject has used anthracyclines and/or taxanes during adjuvant and/or neoadjuvant therapy before breast cancer recurrence. b) The subject has experienced treatment failure during or after chemotherapy based on anthracyclines and/or taxanes. c) According to the investigator's judgment, the Subject is not suitable for anthracyclines and/or taxanes-based chemotherapy as a first-line treatment option.
7. Female subjects are not pregnant, not lactating, and agree to use necessary contraceptive measures.
8. Subjects are able to sign an informed consent form to participate in the study.
9. Have appropriate organ function, as detailed in Table 1; all screening laboratory tests should be completed within 10 days before the start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2028-09-10 (Estimated); Study Completion 2028-09-10 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 24 months
  According to RECIST 1.1 criteria：Disease Progression (PD): Referring to the smallest sum of the diameters of all measured target lesions throughout the entire experimental study, there is a relative increase of at least 20% in the sum of the diameters (if the baseline measurement is the smallest, then the baseline value is used as the reference); in addition, there must be an absolute increase of at least 5 mm in the sum of the diameters (the appearance of one or more new lesions is also considered disease progression).

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China